CLINICAL TRIAL: NCT04631939
Title: Metacognitive Training as a Serious Game: A New Approach for the Treatment of Delusions
Brief Title: Metacognitive Training as a Serious Game
Acronym: Macu'ta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christina Andreou (Other)
Responsible Party: Sponsor-Investigator, Christina Andreou, Principal Investigator, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-02291
Record Dates: First submitted 2020-11-05; First posted 2020-11-17 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia and Related Disorders; Psychotic Disorders; Delusions
Keywords: Psychotic disorders; Delusions; Metacognitive Training; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Delusions

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study intervention (Experimental): The intervention consists of a puzzle adventure game, in which players have to explore the fantasy world "Macu'ta". The puzzles are based on Metacognitive Training for Psychosis (MCT), an intervention using playful, entertaining exercises to increase awareness of reasoning biases in patients and 'sow the seeds of doubt' through corrective ('aha!') experiences. The tasks will address reasoning biases associated with the emergence and maintenance of delusions.
  Interventions: Device: Metacognitive training game
- control intervention (Sham Comparator): The control intervention consists of a puzzles focused exclusively on dexterity and accuracy.
  Interventions: Device: Control games

INTERVENTIONS:
Device: Metacognitive training game — In the fantasy world "Macu'ta", players explore the world by walking around with an avatar in order to find the puzzles and proceed in the game. The intervention consists of 4 different puzzles. Unbeknownst to the player, the first pieces of evidence of each puzzle are often misleading, i.e. indicate the wrong solution, such that hasty decisions are punished. Players receive immediate feedback and are shown the correct response after submitting their solution, as well as explicit cues that educate them on the value of making adequately informed decisions. The order of the puzzles is fixed for each player, but different per session.
  Arms: study intervention
Device: Control games — In the fantasy world "Macu'ta", players explore the world by walking around with an avatar in order to find the puzzles and proceed in the game. The control intervention consists of 4 different puzzle games requiring exclusively dexterity and accuracy (i.e., not including any metacognitive elements). The order of the puzzles is fixed for each player, but different per session.
  Arms: control intervention

SUMMARY:
The project aims to evaluate the efficacy of a therapeutic video game that incorporates elements from metacognitive training on delusions and jumping-to-conclusions in patients with psychotic disorders.

DETAILED DESCRIPTION:
The study is an international, multicenter study and is being conducted in Switzerland (University of Basel) as well as in Germany (University of Lübeck). A total of 36 participants will be included. The estimated duration of the study is 15 months. All participants play a video game from the genre "Third Person Adventure". A character is navigated through a fantasy world using a keyboard and mouse. In the fantasy world, "stations" in the form of glowing gems are sought where players have to solve different tasks.

Participants are randomized to receive either the therapeutic video game with metacognitive training content or another video game with attention and memory tasks ("control intervention"). The control intervention does not include metacognitive tasks. Metacognitive training is an approach for the treatment of psychotic disorders, particularly delusions. The focus of metacognitive training is on thought distortions (so-called "cognitive biases") that are more pronounced in people with psychosis. The control intervention includes easily understandable, playful tasks. The intervention will take 4 appointments within 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 40
* diagnosis of a psychotic disorder and current delusions or a history of delusions

Exclusion Criteria:

* Language skills insufficient for assessments
* IQ < 70
* Secondary psychotic disorders that are clearly induced by general medical conditions or substance use.
* Previous participation in meta-cognitive training for psychosis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change of delusion severity | Change from pre- to post-intervention (4 weeks)
  Item P1 of the Positive and Negative Syndrome Scale (PANSS). Min score = 1, max score = 7, where lower scores indicate better outcome.

SECONDARY OUTCOMES:
Change of total PANSS Score | Change from pre- to post-intervention (4 weeks)
  Total score on the Positive and Negative Syndrome Scale. Lower scores indicate better outcome.
Change of delusional conviction | Change from pre- to post-intervention (4 weeks)
  Total score on the Psychotic Symptom Rating Scales, delusion part (PSYRATS). Lower scores indicate better outcome.
Fish Task: change of number of draws to decision | Change from pre- to post-intervention (4 weeks)
  Number of draws to decision, assessed with the 'Fish task'
Fish Task: change of probability threshold to decision | Change from pre- to post-intervention (4 weeks)
  Probability threshold to decision, assessed with the 'Fish task'

CONTACTS AND LOCATIONS:
Overall Officials: Christina Andreou, PD Dr., Principal Investigator — University of Basel; Stefan Borgwardt, Prof. Dr., Principal Investigator — University of Luebeck
Locations (2):
- Center for Integrative Psychiatry Lübeck, Lübeck, Schleswig-Holstein, Germany
- University Psychiatric Clinics Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All data we will be published on Zenodo under CC0 license.
Supporting Information: Study Protocol
Time Frame: All data will be made openly accessible one year after the study end.
Access Criteria: will be determined at a later time